CLINICAL TRIAL: NCT04480073
Title: Customized CAD/CAM Titanium Meshes for the Guided Bone Regeneration of Severe Alveolar Ridge Defects: Preliminary Results of a Prospective Clinical Follow-up Study in Humans
Brief Title: Guided Bone Regeneration With Customized Titanium Meshes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Matto Chiapasco, Professor, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MChiapasco
Record Dates: First submitted 2020-07-04; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Bone Resorption
Keywords: guided bone regeneration; dental implants; alveolar bone defects; custom-made; Titanium mesh; CAD-CAM; implant-supported prosthesis; autogenous bone
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- edentulous patients with atrophic jaws (Other): patients presenting with severely atrophic edentulous sites in the upper and lower jaw, and requesting implant-supported prosthetic restorations, will be enrolled in this study.
  Interventions: Procedure: Customized CAD-CAM Titanium Mesh (Y-xoss CBR® by Reoss -Filderstadt - Germany) for Guided Bone Regeneration of atrophic alveolar ridges

INTERVENTIONS:
Procedure: Customized CAD-CAM Titanium Mesh (Y-xoss CBR® by Reoss -Filderstadt - Germany) for Guided Bone Regeneration of atrophic alveolar ridges — Step one:1) exposure of atrophic areas; 2) bone harvesting from mandible or calvarium; 3) filling the meshes with a mixture of the autogenous bone and particulated xenograft in a 1:1 ratio; 4) stabilization of the mesh with titanium micro-screws.
  A post-operative cone-beam computed tomography (CBCT) will be done in all patients to have a reference point for the following controls.
  6 months later, patients are re-evaluated with a new CBCT to check bone volumes of the regenerated tissues and to plan implant placement.
  Step two: 1) removal of the meshes; 2) preparation of implant sites (one of which will be randomly chosen to obtain a bone biopsy for histomorphometric analysis); 3) implant placement.
  3 months later, implants will be uncovered and the prosthetic phases will start.
  Patients will be recalled 3, 6, and 12 months later, to assess peri-implant hard and soft tissue conditions, the stability of the reconstructed bone, and the onset of implant-related complications.

SUMMARY:
The aims of this prospective clinical study are to evaluate: a) the effectiveness of digitally customized titanium meshes in association with autologous bone particles and bovine bone mineral and covered with collagen membranes for the regeneration of atrophic edentulous sites; b) the survival rate of implants placed in the reconstructed areas; and c) new bone regeneration from a histomorphometric point of view

DETAILED DESCRIPTION:
Objectives:

* to evaluate the effectiveness of digitally customized titanium meshes for guided bone regeneration with autologous bone chips taken from the mandibular body and/or ramus mixed with bovine bone mineral bone granules (500-1000microns in diameter):

  * complication rate of the reconstructive procedure;
  * assessment of bone gain obtained before implant placement;
* implant survival and implant-related complications 1 year after the starting of prosthetic loading;
* peri-implant bone resorption (MBL) after 1 year from the prosthetic load.
* to perform a histomorphometric analysis of bone samples taken from sites reconstructed according to the principle of Guided Bone regeneration by means of autologous bone chips mixed with a xenograft with a 1:1 ratio and customized titanium mesh.

The following parameters will be analyzed from an histologic point of view:

* bone remodeling and mineralization levels of the new bone matrix
* volumetric tissue fractions
* neo-vascularization

Study method: prospective study - 24 consecutive patients treated (see statistical power analysis)

The study will be performed in accordance with the ISO Standard 14155: 2011, Clinical Investigation of Medical Devices for Human Patients with the Appendices VIII and X of the Medical Device Directive 93/42/ EEC and following the 2004 Helsinki Declaration.

The null hypothesis (H0) is the following: the reconstructed bone is not functionally mature to support implants, masticatory and functional loads after 12 months.

The sample size calculation was performed with the statistical program https://clincalc.com/stats/samplesize.aspx. A literature search on PubMed was performed and revealed that, on average, the percentage of new bone formed after reconstructions with particulate bone autografts and xenografts and titanium mesh is 66% with a standard deviation of 6%. The expected percentage value for the investigator's study was set at 70% with a statistical power of 90% and a two-tier significance level of 0.05.

Data distribution will be analyzed by Shapiro Wilk's normality test, due to the small sample size.

If the data distribution is normal, the comparative analysis for the primary outcome will be performed by T-student test for paired samples. If the data distribution is not normal, a Wilcoxon test will be performed.

The independent variable of the study is the bone reconstruction procedure. The dependent variables are: a) the histomorphometric values of the reconstructed bone; b) the increase (measured in mm) of the bone reconstruction obtained; c) the MBL (in mm) peri-implant 1 year after the prosthetic load.

Data analysis will be performed with SPSS software. Differences will be considered statistically significant for alpha <0.05.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients;
* a minimum age of 18 years;
* relevant or severe bone atrophy at the edentulous sites incompatible with placement of even short (≤6 mm) or narrow (<3 mm) implants in an appropriate and prosthetically guided position;
* adequate compliance of patients, both in terms of oral hygiene and respect the follow-up recalls;
* ability to understand the proposed surgical treatment and to understand and sign the informed consent.

Exclusion Criteria:

* severe kidney and/or liver disease;
* congenital or acquired immunodeficiency;
* ongoing antiblastic chemotherapy at the time of first examination;
* sequelae of radiotherapy in the head and neck area;
* oral mucosa diseases, such as lichen planus;
* full mouth plaque score (FMPS) and full mouth bleeding score (FMBS) < 20%;
* non-compliant patients;
* tobacco abuse (>10 cigarettes per day) or alcohol abuse;
* non compensated diabetes;
* active periodontal disease at the time of first examination ;
* bisphosphonate chemotherapy in progress;
* pregnant women.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Histomorphometric analysis of bone samples taken from the reconstructed sites: bone remodeling and mineralization levels | 6-9 months
  Samples will be processed following a standardized protocol for hard tissues.
  Bone remodeling and mineralization levels of the new bone matrix (expressed in percentage out of the total volume of analyzed sample in cubic mm) will be analyzed from an histologic point of view
Histomorphometric analysis of bone samples taken from the reconstructed sites: Volumetric tissue fractions | 6-9 months
  Samples will be processed following a standardized protocol for hard tissues.
  Volumetric tissue fractions (expressed in percentage out of the total volume of analyzed sample in cubic mm) will be analyzed from an histologic point of view
Histomorphometric analysis of bone samples taken from the reconstructed sites: Neo-vascularization | 6-9 months
  Samples will be processed following a standardized protocol for hard tissues.
  Neo-vascularization (expressed in percentage out of the total volume of analyzed sample in cubic mm) will be analyzed from an histologic point of view
Effectiveness of digitally customized titanium meshes in association with autografts and xenografts for bone regeneration in resorbed jaws: Complication rate of the reconstructive procedure | 6-9 months
  Complication rate of the reconstructive procedure (expressed in percentage and number of patients out of the total) will be analyzed
Effectiveness of digitally customized titanium meshes in association with autografts and xenografts for bone regeneration in resorbed jaws: Assessment of bone gain | 6-9 months
  Assessment of bone gain obtained before implant placement (expressed in mm) will be analyzed
Effectiveness of digitally customized titanium meshes in association with autografts and xenografts for bone regeneration in resorbed jaws: Implant survival | 12 months
  Implant survival (expressed in percentage) will be analyzed
Effectiveness of digitally customized titanium meshes in association with autografts and xenografts for bone regeneration in resorbed jaws: Incidence of implant-related complications | 12 months
  Incidence of implant-related complications 1 year after the starting of prosthetic loading (expressed in percentage) will be analyzed
Effectiveness of digitally customized titanium meshes in association with autografts and xenografts for bone regeneration in resorbed jaws: Peri-implant bone resorption | 6-9 months
  Peri-implant bone resorption (MBL) after 1 year from the prosthetic load (expressed in mm) will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Chiapasco, Professor, Principal Investigator — Department of Biomedical, Surgical and Dental Sciences
Locations (1):
- ASST Santi Paolo e Carlo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
collecting data to verify the effectiveness of bone regeneration with customized titanium meshes and publication of results on peer-reviewed international journals

REFERENCES:
- [Result] Sagheb K, Schiegnitz E, Moergel M, Walter C, Al-Nawas B, Wagner W. Clinical outcome of alveolar ridge augmentation with individualized CAD-CAM-produced titanium mesh. Int J Implant Dent. 2017 Dec;3(1):36. doi: 10.1186/s40729-017-0097-z. Epub 2017 Jul 26. PMID 28748521
- [Result] Seiler M, Kammerer PW, Peetz M, Hartmann A. Customized lattice structure in reconstruction of three-dimensional alveolar defects. Int J Comput Dent. 2018;21(3):261-267. PMID 30264055
- [Result] Sumida T, Otawa N, Kamata YU, Kamakura S, Mtsushita T, Kitagaki H, Mori S, Sasaki K, Fujibayashi S, Takemoto M, Yamaguchi A, Sohmura T, Nakamura T, Mori Y. Custom-made titanium devices as membranes for bone augmentation in implant treatment: Clinical application and the comparison with conventional titanium mesh. J Craniomaxillofac Surg. 2015 Dec;43(10):2183-8. doi: 10.1016/j.jcms.2015.10.020. Epub 2015 Oct 23. PMID 26603108